CLINICAL TRIAL: NCT05451667
Title: A Phase I, Randomized, Double-Blind, Placebo Controlled Single-Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Topical Application of YJ001 in Healthy Volunteers
Brief Title: Single-Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of YJ001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuejia Pharmaceuticals (USA), Inc. (Industry)
Collaborators: Zhejiang Yuejia Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zhejiang Yuejia Pharmaceuticals Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YJ001-102
Record Dates: First submitted 2022-06-28; First posted 2022-07-11 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Safety and Tolerability
MeSH Terms: interventions — Hypromellose Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded with regard to the study treatment that subjects receive, without the Investigator, the Sponsor, or the subjects being aware of whether YJ001 or the placebo is administered. All decisions concerning dose escalation will be made in a blinded manner by the safety review committee (SRC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (6 active, 2 placebo) (Experimental): 148 mg
  Interventions: Drug: YJ001 for Spray Use; Drug: Placebo of YJ001 for Spray Use
- Cohort 2 (6 active, 2 placebo) (Experimental): 296 mg
  Interventions: Drug: YJ001 for Spray Use; Drug: Placebo of YJ001 for Spray Use
- Cohort 3 (6 active, 2 placebo) (Experimental): 552 mg
  Interventions: Drug: YJ001 for Spray Use; Drug: Placebo of YJ001 for Spray Use
- Cohort 4 (6 active, 2 placebo) (Experimental): 828 mg
  Interventions: Drug: YJ001 for Spray Use; Drug: Placebo of YJ001 for Spray Use

INTERVENTIONS:
Drug: YJ001 for Spray Use — YJ001 (active ingredient)
  Other Names: YJ001
Drug: Placebo of YJ001 for Spray Use — Hydroxypropyl Methylcellulose
  Other Names: Hydroxypropyl Methylcellulose

SUMMARY:
This phase I, randomized, double-blind, placebo controlled study is to investigate the safety, tolerability and pharmacokinetics (PK) of topically administered YJ001 in a single-ascending dose (SAD) fashion in healthy volunteers between 18 to 55 years of age, to establish the dosage range for spray use, and to provide a dosage regimen for Phase I multiple-ascending dose (MAD) study in healthy subjects. The study is to enroll 4 cohorts, the doses of which are 148, 296, 552 and 828 mg, with the option to enroll 2 additional cohorts (8 subjects for each cohort) without requiring a protocol amendment. Subjects will be screened between Day -28 and Day -2 and will be admitted to the clinic on Day -1. Subjects will be housed within the clinic from Day -1 through Day 8 and will be discharged on Day 8 after all scheduled study procedures have been completed.

DETAILED DESCRIPTION:
This phase I, randomized, double-blind, placebo controlled study is to investigate the safety, tolerability and pharmacokinetics (PK) of topically administered YJ001 in a single-ascending dose (SAD) fashion in healthy volunteers between 18 to 55 years of age, to establish the dosage range for spray use, and to provide a dosage regimen for Phase I multiple-ascending dose (MAD) study in healthy subjects. The study is to enroll 4 cohorts, the doses of which are 148, 296, 552 and 828 mg, with the option to enroll 2 additional cohorts (8 subjects for each cohort) without requiring a protocol amendment. Each cohort will consist of 8 subjects (6 active; 2 placebo). Each subject will be administered a single dose of YJ001 as multiple sprays (8 sprays/foot for Cohort 1, 16 sprays/foot for Cohort 2, 16 sprays/foot for Cohort 3, and 24 sprays/foot for Cohort 4) topically on both feet; and below the ankle, with the administration area set as 450 cm2 (both feet).

Safety will be evaluated by assessing incidence and severity of adverse events (AEs) and serious adverse events (SAEs); observed values and changes in baseline of clinical safety laboratory test results, 12-lead electrocardiogram (ECG), vital signs; and physical examination inclusive of skin reaction findings at the Investigational Product (IP) administration sites.

For pharmacokinetics evaluation, serial blood samples will be collected in the subjects of Cohorts 2 to 4 for up to 7 days following a single dose to assess the PK of YJ001 and metabolites in plasma. Pooled urine samples will be collected in the subjects of Cohorts 2 to 4 to evaluate renal excretion of YJ001 and metabolites.

Subjects will be screened between Day -28 and Day -2 and will be admitted to the clinic on Day -1. Subjects will be housed within the clinic from Day -1 through Day 8 and will be discharged on Day 8 after all scheduled study procedures have been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between the ages of 18-55 years at screening, both inclusive.
2. Subjects voluntarily consenting for participation in the study and have signed informed consent document. Subjects are required to understand verbal and/or written English or any other language in which a certified translation of the informed consent is available.
3. The body weight of male and female should be ≥ 50.0 and ≥ 45.0 kg, respectively; have a body mass index (BMI) between 19.0 to 32.0 kg/m2 (both inclusive) at screening, calculated as weight (kg)/height2 (m2). Subjects must have two feet. Each foot must have five digits. Each foot must have at least total surface area of 450 cm2 measured from below the ankle to the toes including both dorsum and plantar areas.
4. Medical history without any clinically significant pathology/surgery in the last 6 months.
5. Resting supine blood pressure 90-140 (systolic)/60-90 (diastolic) mmHg, a resting pulse rate of 45-100 beats per minute at screening.
6. Calculated creatinine clearance should be within the normal range using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Based Equation1.
7. Computerized 12-lead ECG recording without signs of clinically significant pathology or showing no clinically significant deviation as judged by the Investigator at screening and pre-dose.
8. Subjects with either C-reactive protein of up to 3.0 mg/L or Hemoglobin A1C of up to 5.9%.
9. Males must not to donate sperm until 90 days after last dose of study drug and must be willing to use a condom during heterosexual activity for up to 90 days after the application of the study drug.
10. Females must be either postmenopausal for at least 1 year, surgically sterile (bilateral tubal ligation [including clip, cauterization methods and coil], bilateral oophorectomy or hysterectomy, and needs to be confirmed follicle stimulating hormone [FSH] level >40 IU/L), or of childbearing potential either practicing true abstinence or practicing 2 effective means of contraception for 3 weeks prior to study drug administration, and until 28 days after study drug administration:

    1. Intrauterine device (IUD) or IUD hormone-releasing system.
    2. Combined estrogen and progestogen containing hormonal contraception (oral, intravaginal, or transdermal) associated with inhibition of ovulation.
    3. Progesterone-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation.
    4. Intrauterine hormone-releasing system.
    5. Double-barrier method (condoms, contraceptive sponge, diaphragm, or vaginal ring with spermicide).
11. All values of hematology and biochemistry of blood and urine are within allowed normal limits or not clinically significant as judged by the Investigator.
12. Able and willing to comply with all study requirements.

Exclusion Criteria:

1. Current participation in another investigational drug or device study or treated with an investigational drug within 30 days or 5 half-lives, whichever is longer, before dosing.
2. History/evidence of clinically relevant pathology related to cardiovascular (CVS), central nervous system (CNS), respiratory tract, gastrointestinal (GI), endocrinology, immunology, hematology, or any other systemic disorder/major surgeries within the last 6 months that in the opinion of the Investigator would confound subject's participation and follow-up in the clinical trial.
3. History of clinically significant drug, food allergy, skin allergy, or sensitivity to drugs of the same class (e.g., 5-aminosalicylic acid, sulfasalazine, and salicylates) or known hypersensitivity to YJ001 or any of its components.
4. History of asthma. Adults with history of benign (resolved) childhood asthma may be included.
5. Consumed more than 28 units of ethanol per week at any time in the 6 months before dosing (1 unit of ethanol is equivalent to 12 ounces of beer, 5 ounces of wine, or 1.5 ounces of spirits) or history of drug or alcohol abuse within the 6 months or evidence of such abuse as indicated by inquiry, medical history or the laboratory assays conducted during screening.
6. Positive screening or check-in alcohol/drugs of abuse/cotinine screen.
7. Positive test results for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Screening. SARS-CoV-2 testing will be either NP or nasal swab PCR performed at Day -4, and in accordance with Centers for Disease Control and Prevention (CDC), FDA and local health authorities at the time of enrollment for this study. Participants not willing to comply with Pharmaron's COVID 19 policy.
8. Female volunteers who are pregnant or lactating.
9. Systemic or topical use of aspirin or salicylic acid containing products or sulfasalazine/salicylic acid derivatives within 14 days of study drug dosing.
10. Use of other prescription and non-prescription medications (with the exception of oral contraceptives, combined estrogen and progestogen containing hormonal contraception and progestogen-only hormonal contraception), including nonsteroidal anti-inflammatory drugs, NSAIDs (i.e., ibuprofen), blood thinners, or sucralfate or herbal preparations within 14 days or 5 half-lives (whichever is longer) before study drug dosing, or use of an over-the-counter medication, vitamins, or supplements (including fish liver oils) within 14 days before study drug dosing.
11. Any subject who has received any known hepatic or renal clearance (CLr) altering agents (e.g., erythromycin, cimetidine, barbiturates, phenothiazines, or herbal/plant-derived preparations such as St. John's Wort, etc.) for a period of 30 days prior to the dose of study medication.
12. Positive screen on Hepatitis B, Hepatitis C, or Human immunodeficiency virus (HIV) at the time of screening evaluations.
13. Unwilling to stay in the clinical unit for the required duration as per the protocol or consume the standard meal to be provided as per the protocol.
14. History of blood donation of more than 500 mL in the last 2 months prior to screening.
15. Consumption of xanthine containing food or beverages (like tea, coffee, chocolates, or cola drinks) 24 hours prior to dosing.
16. Any subject who consumes more than 5 cigarettes per day within 30 days before study drug dosing or who cannot stop using any tobacco- or nicotine-containing product during the duration of the trial.
17. History or evidence of poor venous access.
18. History of bleeding disorders.
19. Any other medical, psychological, or social condition which, in the opinion of the Investigator, would prevent the subject from fully participating in the study, would represent a concern for study compliance, or would constitute a safety concern to the subject.
20. Presence of skin disorders, tattoos, or other skin conditions on either foot that may interfere with the objectives of the study (as per investigator evaluation).
21. Use of any kind of topical lotions on the feet for 72 hours prior to the study that may interfere with the objectives of the study (as per investigator evaluation).
22. An employee of the study center or Sponsor or family member of a study center employee.
23. Have a significant acute illness within 7 days prior to study drug administration or have had a major illness or hospitalization within 1 month prior to study drug administration.
24. Any subject considering or scheduled to undergo any surgical procedure from screening to follow-up visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and significant laboratory abnormality | Day -28 to Day 8
  If ≥ 2 subjects assigned to YJ001 in a cohort experience any of the following:
  1. A Grade ≥ 2 adverse event.
  2. A Grade ≥ 2 clinically significant laboratory abnormality.
Systemic exposure of the 4 analytes to be assayed | Day 1 to Day 8
  If ≥ 1 subject meets/exceeds the exposure limits for any of YJ001 and its metabolites (YJ001-A, YJ001-B, and/or YJ001-C) or if subjects are expected to exceed the specific exposure limits for any analyte at a next planned dose level.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No